CLINICAL TRIAL: NCT01954316
Title: An Open Label, Dose Escalation, Safety, and Pharmacokinetic Study of CFI-400945 Fumarate Administered Orally to Patients With Advanced Cancer
Brief Title: A Study of CFI-400945 Fumarate in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Princess Margaret Cancer Foundation (Other); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CFI-400945-CL-001
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Advanced Cancer
Keywords: advanced cancer; CFI-400945 fumarate; polo-like kinase 4; PLK4; tablet; dose escalation; genetic testing
MeSH Terms: interventions — 2-(3-(4-((2,6-dimethylmorpholino)methyl)styryl)-1H-indazol-6-yl)-5'-methoxyspiro(cyclopropane-1,3'-indolin)-2'-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CFI-400945 fumarate Schedule A (Experimental): CFI-400945 fumarate tablets daily dosing expansion at 64mg
  Interventions: Drug: CFI-400945
- CFI-400945 fumarate Schedule B (Experimental): CFI-400945 fumarate tablets intermittent dosing schedule, 2 days on/5 days off. Escalation at following levels: 96mg, 128mg
  Interventions: Drug: CFI-400945
- CFI-400945 fumarate Schedule C (Experimental): CFI-400945 fumarate tablets intermittent dosing schedule, 1 day on/6 days off. Escalation will start at MTD of Schedule B
  Interventions: Drug: CFI-400945

INTERVENTIONS:
Drug: CFI-400945 — Polo-like kinase 4 (PLK4) inhibitor

SUMMARY:
This is a phase 1 study to test different doses of a new investigational drug called CFI-400945 to see which dose is safer in people. This study will also look at the safety of CFI-400945 and to study its effects on patients with advanced cancers. This drug has been tested in animals but not yet in people.

CFI-400945 is an oral (taken by mouth) drug that works by blocking polo-like kinase 4 (PLK4) from working. PLK4 is a protein that is important in regulating cell growth and division and cell death. Many tumors are shown to make too much PLK4. When there is too much PLK4 produced, it is believed to lead to uncontrolled cancer cell growth and division. Therefore, by blocking this protein from working, it is believed to stop tumors growing or shrink them.

DETAILED DESCRIPTION:
All participants will receive CFI-400945. At the beginning of the study, participants are given a low dose of CFI-400945 and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then more participants are asked to join the study and are given a higher dose of study drug. Participants joining the study later on will get higher doses of study drug than participants who join earlier. This will continue until the highest dose of study drug that can be taken without severe side effects is found (called maximum tolerated dose). Doses higher than that will not be given.

After the best dose of study drug is found, additional participants will be asked to join the study and will be given the study drug at the maximum tolerated dose to further test the safety and the drug at that dose.

ELIGIBILITY:
Inclusion Criteria:

* Have histologic or cytological proof of advanced cancer that has progressed and for which there is no further standard anticancer therapy available in the opinion of the investigator.
* Patients must have measurable disease as per RECIST v1.1
* Are 18 years of age or older.
* Have clinically acceptable laboratory screening results within certain limits
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Able to swallow oral medications.
* Have a life expectancy greater than 3 months.
* Women and men of child producing potential must agree to use highly effective means of contraception during study participation, and for at least 30 days after the last administration of study medication.
* Negative serum pregnancy test with 72 hours prior to start of study drug
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Have received radiotherapy, chemotherapy, biological therapy or investigational treatment less than four weeks (six weeks for nitrosourea or mitomycin C) prior to first dose of study medication or have not recovered from all acute toxicities from prior treatments.
* Patients who have received growth factors within 14 days prior to initiation of dosing of CFI-400945 fumarate.
* Have active, acute, or chronic clinically significant infections.
* Have uncontrolled severe hypertension
* Have clinical symptomatic congestive heart failure defined at >= Class II of the New York Heart Association functional classification system or LVEF < 50% at baseline.
* Have active angina pectoris or recent myocardial infarction (within 6 months).
* Have chronic atrial fibrillation or QTc of greater than 470 msec, as calculated by Bazett's correction formula.
* Have had major surgery within 21 days of starting therapy. Placement of a venous access device within 21 days of starting therapy is allowed.
* Have additional uncontrolled serious medical or psychiatric illness.
* Have any medical condition that could impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting.
* Known central nervous system metastasis. Patients with history of central nervous system metastases are eligible if they are clinically or radiographically stable for at least 3 months and not taking steroids or anticonvulsants.
* Patients being treated with full dose warfarin are excluded. Patients with history of deep vein thrombosis or pulmonary embolus who are being treated with therapeutic doses of low molecular weight heparin or prophylactic dose anticoagulants may be enrolled.
* Patients being treated with certain drugs not acceptable while receiving CFI-400945 fumarate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03; Primary Completion 2021-07 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Highest dose level that does not lead to unacceptable toxicity in two or more patients in a dosing group over a range of doses and schedules | From first dose of study drug until the date of unacceptable toxicity, throughout the study completion, up to 2 years
  Though evaluation of AEs and DLTS of all patients who have received study drug

SECONDARY OUTCOMES:
Pharmacokinetic profile of CFI-400945 fumarate (please see description below) over a range of doses and schedules | Day 1 and Day 28 of Cycle 1 prior to first dose and at 0.5, 1, 2 (± 5 minutes), 4, 6, 8, 10-12 (± 15 minutes), and 24 hours (± 60 minutes) following dosing. Day 1 of Cycle 2 and future cycles, prior to dosing.
  * Area under the plasma concentration-time curve (AUC)
  * Elimination half-life (T½)
  * Maximum plasma concentration (Cmax)
  * Minimum plasma concentration (Cmin)
  * Time when Cmax occurs (Tmax)
  * Average plasma concentration at steady state (Cavg)
Number of patients with evidence of benefit over a range of doses and schedules | through study completion, up to 2 years
  response to treatment and/or clinical benefit or tumor marker improvement
Number of side effects occurring and severity | through study completion, up to 2 years
  by frequency and severity of treatment emergent adverse events in cancer patients
Evaluate the genomic alterations and other molecular features which are associated with response and/or clinical benefit with CFI-400945-CL fumarate treatment | At any time from when the patient reaches 3 months on trial or more at the time of progression
  Through optional tumor biopsies; Gene or protein expression levels
to evaluate pharmacodynamics effects relative to CFI-400945 fumarate at MTD | At any time from when the patient reaches 3 months on trial or more at the time of progression, up to two years
  Through baseline biopsy comparisons with optional tumor biopsy at the time of progression
Determine evidence of benefit in cancer patients when CFI-400945 fumarate is administered orally at the MTD (expansion) | At any time from when the patient reaches 3 months on trial or more at the time of progression, up to two years
  Evaluating tumor response(if appropriate) and/or clinical benefit or tumor marker improvement
To evaluate possible mechanisms of resistance to CFI-400945 fumarate at MTD | At any time from when the patient reaches 3 months on trial or more at the time of progression, up to two years
  Through optional baseline biopsy comparisons with optional tumor biopsy at the time of progression
Determine recommended Phase 2 dose for CFI-400945 fumarate | Based on safety profile evaluated throughout the DLT period, which is Cycle 1 (each cycle being 28 days) of treatment, and through study completion up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (2):
- UCLA Medical Center, Santa Monica, California, United States
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Veitch ZW, Cescon DW, Denny T, Yonemoto LM, Fletcher G, Brokx R, Sampson P, Li SW, Pugh TJ, Bruce J, Bray MR, Slamon DJ, Mak TW, Wainberg ZA, Bedard PL. Safety and tolerability of CFI-400945, a first-in-class, selective PLK4 inhibitor in advanced solid tumours: a phase 1 dose-escalation trial. Br J Cancer. 2019 Aug;121(4):318-324. doi: 10.1038/s41416-019-0517-3. Epub 2019 Jul 15. PMID 31303643
- See also: Jacqueline Mason et al. Functional characterization of CFI-400945, a Polo-like kinase 4 inhibitor, as a potential anticancer agent. Cancer Cell. 2014 Aug 11;26(2):163-76. — https://doi.org/10.1016/j.ccr.2014.05.006